CLINICAL TRIAL: NCT01519505
Title: Diabetes in Europe - Prevention Using Lifestyle, Physical Activity and Nutritional Intervention in Catalonia(DE-PLAN-CAT).
Brief Title: Diabetes in Europe - Prevention Using Lifestyle, Physical Activity and Nutritional Intervention in Catalonia
Acronym: DE-PLAN-CAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05/38
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Prevention; Diabetes mellitus; Lifestyle changes; Cardiovascular risk; Cost-effectiveness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Complete lifestyle counseling including
  1. Individual intervention, OR
  2. Group intervention
  Interventions: Behavioral: Lifestyle intervention
- Usual health care (No Intervention): Usual health care, including self-administered information by leaflets

INTERVENTIONS:
Behavioral: Lifestyle intervention — INDIVIDUAL INTERVENTIONS They were programmed to come the nurse office three times (1 ½ -2 hours each). Individual intervention efforts outside of weight control and other intervention groups were also supported. In fact, this kind of intervention was similar to the group intervention but one-by-one participant subject. GROUP INTERVENTIONS Six-hour educational programme structured in 2 to 4 sessions with 5 to 15 participants. We called all participants to remind them their group schedule (date/hour). The methods used in the group intervention were variable depending on the experience of the manager, group member' s needs and skills available (empowerment). Results were based on motivation, support from the other members, peer support and positive feedback.
  Other Names: Individual intervention; Group intervention
  Arms: Lifestyle counseling

SUMMARY:
Public health strategy on type2 diabetes prevention in primary health care. European coordinated project (DE-PLAN) adapted to Catalonia (DE-PLAN-CAT). Two-step multicentre cohort study: cross-over period (screening) plus a follow-up period (preventive intervention): 12 centres, 7 working-groups, 42 units, 106 professionals). Interventions: Randomized non-invasive diabetes screening program by means of the FINDRISC score comparing with the oral glucose tolerance test results. At least one third of the screened subjects is expected to present high-risk criteria. They will choose 1 out of 3 interventions to modify lifestyle: self-acting vs. individualized or group-based educative (6-hour, 3 or 4 sessions program). Participants' motivation will be periodically reinforced. Follow-up will be focused on diabetes incidence, cardiovascular risk (HearthScore, Regicor scores), lifestyle-quality of life (assessed by European peer-reviewed questionnaires) and cost-effectiveness analysis. First-year results includes: protocol, measurement tools and database available, screening concluded (n=2082) and European intervention manual on type 2 diabetes prevention started.

DETAILED DESCRIPTION:
Diabetes is one of the most devastating diseases because of its big impact on public health. Taking fast decisions and vigorous actions like the ones proposed by this European project (DE-PLAN) adapted to the Spanish and the Catalan actual situation (coordinated project FIS and DE-PLAN-CAT respectively) can avert it.

We consider a two-step strategy whose main objective is the primary prevention of diabetes in the European population at highest-risk. At the first stage, a non-invasive screening program will evaluate the risk of diabetes by means of a validated questionnaire (FINDRISK survey). It will be distributed at random to 2000 outpatients of public health service in Catalonia. It involves twenty primary care facilities that refer to five different centers where research scientists (executive committee) are coordinated by the head of these centers (coordinating committee) and are organised (managing committee) according to the European regulation (central committee). One third of the subjects are expected to present high-risk criteria. They will choose one out of three possible interventions to modify their lifestyle (informative approach, one-to-one or group training). For the last options, a 6-hour training program will be carried out in four sessions lasting 1,5 hours each. The trainers in charge will periodically stimulate the participants motivation.

The study will go on in the routine health care and it will assess diabetes incidence according to the economic estimation of the cost-effectiveness relation of the adopted measures involved in health care policies and prevention programs.

This project aims to evidence how the already known efficacy of these types of programs can apply to its effectiveness (on large populations) and its cost-effectiveness (in socio-economic terms). Other objectives are 1) to create one bigger database of diabetes and cardiovascular disease risks and 2) to contribute to the edition of a European manual on type 2 diabetes prevention.

ELIGIBILITY:
Inclusion Criteria:

* High risk (> or equal 14 points in FINDRISC score)
* PTOG with IFG/ITG or both
* Able to sign informed consent

Exclusion Criteria:

* Type 2 diabetes in screening
* Low risk (< 14 points in FINDRISC)
* Terminal diseases

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2082 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Incident cases of type 2 diabetes | 4 years
  New cases of type 2 diabetes in subjects with high risk during the duration of the study

SECONDARY OUTCOMES:
Evaluation of quality of life | 4 years
  Quality of life in the 15-D questionnaire
Cost-effectiveness | 4 years
  Evaluation of cost-effectiveness of the efforts to prevent one case of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Costa, MD PhD, Principal Investigator — Catalan Institute of Health
Locations (1):
- IDIAP Jordi Gol, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Costa B, Barrio F, Cabre JJ, Pinol JL, Cos X, Sole C, Bolibar B, Basora J, Castell C, Sola-Morales O, Salas-Salvado J, Lindstrom J, Tuomilehto J; DE-PLAN-CAT Research Group. Delaying progression to type 2 diabetes among high-risk Spanish individuals is feasible in real-life primary healthcare settings using intensive lifestyle intervention. Diabetologia. 2012 May;55(5):1319-28. doi: 10.1007/s00125-012-2492-6. Epub 2012 Feb 10. PMID 22322921